CLINICAL TRIAL: NCT02372526
Title: The Effect of Different Macronutrients on Gastrointestinal Hormone Secretion After Gastric Bypass Operation
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kirstine Nyvold Bojsen-Moeller (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Sponsor-Investigator, Kirstine Nyvold Bojsen-Moeller, Postdoc, Hvidovre University Hospital
Organization: Hvidovre University Hospital (Other)
Other Study IDs: CZJ-MA-14
Record Dates: First submitted 2015-02-20; First posted 2015-02-26 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Bariatric Surgery (Gastric Bypass); Overweight
Keywords: Glucagon-like Peptide-1; Glucose-dependent insulinotropic peptide; Glucagon; Peptide YY 3-36; Ghrelin; Body Weight; Obesity; Overnutrition; Overweight; Gastrointestinal Agents; GLP-1 secretagogue
MeSH Terms: conditions — Overweight; Body Weight; Obesity; Overnutrition | interventions — CD36 Antigens

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma and serum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 10 Roux-en-Y gastric bypass patients: Isocaloric amounts of specific macronutrients is mixed with 4 g vegetable bouillon and tested against each others ability to induce GLP-1 secretion. The mealtest takes place at 4 different days with 3-14 days separation.
  Interventions: Other: Mealtest: High protein 200 kcal 200 ml liquid meal consumed during 10 minutes; Other: Mealtest: High fat 200 kcal 200 ml liquid meal consumed during 10 minutes; Other: Mealtest: High carbohydrate 200 kcal 200 ml liquid meal consumed during 10 minutes; Other: Mealtest: High fat 200 kcal 200 ml liquid meal with pancreatic lipase inhibitor consumed during 10 minutes
- 10 Healthy Control subjects: Isocaloric amounts of specific macronutrients is mixed with 4 g vegetable bouillon and tested against each others ability to induce GLP-1 secretion. The mealtest takes place at 4 different days with 3-14 days separation.
  Interventions: Other: Mealtest: High protein 200 kcal 200 ml liquid meal consumed during 10 minutes; Other: Mealtest: High fat 200 kcal 200 ml liquid meal consumed during 10 minutes; Other: Mealtest: High carbohydrate 200 kcal 200 ml liquid meal consumed during 10 minutes; Other: Mealtest: High fat 200 kcal 200 ml liquid meal with pancreatic lipase inhibitor consumed during 10 minutes

INTERVENTIONS:
Other: Mealtest: High protein 200 kcal 200 ml liquid meal consumed during 10 minutes
  Other Names: LACPRODAN SP-9225 INSTANT Whey Protein Isolate
Other: Mealtest: High fat 200 kcal 200 ml liquid meal consumed during 10 minutes
  Other Names: Lurpak® smør(butter) 81% fat
Other: Mealtest: High carbohydrate 200 kcal 200 ml liquid meal consumed during 10 minutes
  Other Names: Urtegaarden Druesukker (Dextrose monohydrat)
Other: Mealtest: High fat 200 kcal 200 ml liquid meal with pancreatic lipase inhibitor consumed during 10 minutes
  Other Names: Lurpak® smør(butter) 81% fat with 120 mg Xenical® Orlistat

SUMMARY:
The purpose of this study is to determine the type of macronutrient (carbohydrate, lipid or protein) that most potently stimulates the endogen secretion of different gut hormones (primary outcome = Glucagon-Like peptide-1) in gastric bypass operated patients. The study also includes a comparison of the secretion of gut hormones after oral intake of lipid with or without a pancreatic lipase inhibitor.

ELIGIBILITY:
RYGB Patients:

Inclusion Criteria:

* Underwent RYGB surgery more than 18 months earlier, weight stabile (+/- 5 kg during 1 month)

Exclusion Criteria:

* Inadequate thyroid substitution, undergoing treatment with drugs known to interact with Orlistat (such as cyclosporine, anticoagulating agents, amiodarone, amlodipine and epileptics), where pausing the treatment with these is not an option. Type 1 or 2 diabetes mellitus now or prior to RYGB operation. Serious heart or respiratory illness. Haemoglobin levels below 6,5 mM.

Healthy control subjects:

Inclusion Criteria:

* Have not underwent bariatric surgery.

Exclusion Criteria:

* Inadequate thyroid substitution, undergoing treatment with drugs known to interact with Orlistat (such as cyclosporine, anticoagulating agents, amiodarone, amlodipine and epileptics), where pausing the treatment with these is not an option. Type 1 or 2 diabetes mellitus now or prior. Serious heart or respiratory illness. Haemoglobin levels below 6,5 mM.

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: RYGB Patients who have underwent RYGB surgery more than 18 months earlier, weight stabile (+/- 5 kg during 1 month). Healthy control subjects who have not underwent bariatric surgery.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2015-01; Primary Completion 2016-08 (Actual); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Within group difference in Glucagon-like Peptide 1 secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
  I.e. Comparison of GLP-1 secretion (iAUC) as a result of intake of different macronutrients between a) gastric bypass patients only b) healthy volunteers only.

SECONDARY OUTCOMES:
Within group difference in Glucagon secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Within group difference in Glucose-dependent insulinotropic peptide secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Within group difference in Cholecystokinin secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Within group difference in Peptide YY 3-36 secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Within group difference in Ghrelin secretion (evaluated by iAUC). | 0, 30, 45, 60, 120, 180, 240
Within group difference in Changes in bile acids. | 0, 30, 45, 60, 120, 180, 240
Within group difference in Changes in glycerol, triacylglycerol and free fatty acids. | 0, 30, 45, 60, 120, 180, 240
Within group difference in Insulin secretion (evaluated by iAUC). | 2xBasline, 0, 10, 15, 20, 30, 40, 45, 60, 90, 120, 180, 240
Within group difference in Plasma glucose concentration. | 2xBasline, 0, 5, 10, 15, 20, 25, 30, 40, 45, 60, 90, 120, 180, 240
Within group difference in Visual Analog Scale. | 0, 30, 60, 90, 120, 180, 240
  Hunger, satiety, abdominal pain and nausea measured by standard 10 cm Visual Analog Scale
Within group difference in Ad libitum food intake (grams). | 240
Within group difference in Heart rate (bpm). | 2xBasline, 0, 5, 10, 15, 20, 25, 30, 40, 45, 60, 90, 120, 180, 240
Within group difference in Blood pressure (mmhg). | 0, 15, 30, 45, 60, 90, 120, 180, 240

OTHER OUTCOMES:
Between groups difference in Glucagon-like Peptide 1 secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
  I.e. Comparison of GLP-1 secretion (iAUC) as a result of intake of different macronutrients between Gastric bypass operated patients and Healthy volunteers.
Between groups difference in Glucagon secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Between groups difference in Glucose-dependent insulinotropic peptide secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Between groups difference in Cholecystokinin secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Between groups difference in Peptide YY 3-36 secretion (evaluated by iAUC). | Basline, 0, 15, 30, 45, 60, 90, 120, 180, 240
Between groups difference in Ghrelin secretion (evaluated by iAUC). | 0, 30, 45, 60, 120, 180, 240
Between groups difference in Changes in bile acids. | 0, 30, 45, 60, 120, 180, 240
Between groups difference in Changes in glycerol, triacylglycerol and free fatty acids. | 0, 30, 45, 60, 120, 180, 240
Between groups difference in Insulin secretion (evaluated by iAUC). | 2xBasline, 0, 10, 15, 20, 30, 40, 45, 60, 90, 120, 180, 240
Between groups difference in Plasma glucose concentration. | 2xBasline, 0, 5, 10, 15, 20, 25, 30, 40, 45, 60, 90, 120, 180, 240
Between groups difference in Visual Analog Scale. | 0, 30, 60, 90, 120, 180, 240
  Hunger, satiety, abdominal pain and nausea measured by standard 10 cm Visual Analog Scale
Between groups difference in Ad libitum food intake (grams). | 240
Between groups difference in Heart rate (bpm). | 2xBasline, 0, 5, 10, 15, 20, 25, 30, 40, 45, 60, 90, 120, 180, 240
Between groups difference in Blood pressure (mmhg). | 0, 15, 30, 45, 60, 90, 120, 180, 240

CONTACTS AND LOCATIONS:
Locations (1):
- Endocrinology Research Center, Hvidovre University Hospital, Hvidovre, Copenhagen, Denmark